CLINICAL TRIAL: NCT03765515
Title: A Prospective, Randomized, Multi-Center Clinical Study to Evaluate the Safety and Efficacy of Q-Fix All-Suture Anchor in Arthroscopic Repair of Shoulder Soft Tissue in Chinese Patients
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Q-Fix Trial in Chinese Patients
Acronym: Q-Fix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-5010-05
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Arthroscopy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Q-Fix (Experimental): Q-Fix has the advantages of all-suture implant and has the same or better performance than the traditional anchor.
  * Consistent activation effect
  * Excellent performance
  * Streamlined technique Q-fix is an experimental Arm.
  Interventions: Device: Q-Fix
- Twinfix Ti (Active Comparator): The Smith & Nephew's marketed Twinfix Suture Anchor is selected as the control product. This product is composed of anchor, suture, suture needle and inserter. The anchor is made of Ti6Al4V titanium alloy conforming to ISO5832-3. The Durabraid suture is made of polyester (Polyethylene terephthalate) conforming to YY 0167. Ultrabraid suture is made of two materials of UHMWPE and polypropylene monofilaments conforming to GB/T 19701.1. The suture needle is made of Type 420B stainless steel conforming to YY/T 0726. The stem portion of inserter that comes into contact with the body is made of Type 630B stainless steel conforming to YY/T 0726.
  Interventions: Device: Twinfix Ti

INTERVENTIONS:
Device: Twinfix Ti — The purpose is to evaluate the safety and efficacy of Q-Fix in patients requiring the repair of soft tissue of shoulder who receive the arthroscopic repair of soft tissue using Q-Fix, when compared with the patients receiving the treatment with Twinfix Ti Suture Anchor. The result of this trial will be used for the Q-Fix All-suture Anchor registration in China.
  Arms: Twinfix Ti
Device: Q-Fix — Q-Fix
  Arms: Q-Fix

SUMMARY:
Protocol synopsis Title of Study: A Prospective, Randomized, Multi-Center Clinical Study to Evaluate the Safety and Efficacy of Q-Fix All-Suture Anchor in Arthroscopic Repair of Shoulder Soft Tissue in Chinese Patients

Study Design: Prospective, multicenter, comparative, randomized, concurrent control Study Type: Randomized Controlled Trial (RCT) Study Product: Q-Fix All-Suture Anchor Comparison Group Twinfix Ti Suture Anchor Study Purpose: The purpose of this study is to evaluate the safety and efficacy of Q-Fix All-suture Anchor in patients requiring the repair of soft tissue of shoulder who receive the arthroscopic repair of soft tissue using Q-Fix All-suture Anchor, when compared with the patients receiving the treatment with Twinfix Ti Suture Anchor. The result of this trial will be used for the Q-Fix All-suture Anchor registration in China.

Primary Objective: The primary objective of this study is to confirm that the clinical outcome of subjects receiving the treatment with Q-Fix All-suture Anchor is non-inferior to that of the subjects receiving the treatment with Twinfix Ti Suture Anchor during the same period, at 6 months after the repair of soft tissue of shoulder, taking the mean Constant score as efficacy endpoint.

Secondary Objective(s): The secondary objective of this study is to determine the safety and efficacy of Q-Fix All-suture Anchor at 12 months after repair of soft tissue of shoulder.

Statistical Rationale: The primary efficacy endpoint of this study is Constant score at 6 months after operation. The non-inferiority testing is performed for efficiency of primary efficacy endpoint; the test hypothesis is as follows:

Invalid hypothesis: H0: μ1-μ2 ≤ -δ Alternative hypothesis: H1: μ1-μ2 > -δ Where, μ1 and μ2 are the mean Constant scores in the test and control group, respectively. δ is the non-inferiority margin, which is set to 10. The hypothesis will be tested by two-sided t-test at the alpha level of α=0.025 (one-tailed test). the A non-inferior test will be conducted on the Constant scores in the test and control groups. The 95% confidence interval for the difference between two groups will be calculated. If the lower limit of 95%CI for the efficiency difference between two groups is greater than -9, it is considered that the test group is non-inferior to the control group.

Sample Size: 128 (64 in each group) Number of Study Sites: Approximate 5 clinical sites Targeted Global Regions: China

DETAILED DESCRIPTION:
Study Duration: 24 months = 12 months of recruitment + 12 months of follow up (From the start of screening to the time that the last subject completes the trial) Primary endpoint: Constant score at 6 months after operation for the shoulder Secondary endpoint(s): ASES score Rowe score WORC questionnaire Incidence of rotator cuff re-tear Recurrence rate of shoulder joint instability Anchor pullout rate Adverse event Radiographic evaluation results Constant score Safety Data AEs, SAEs, ADEs, UADEs

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 18 - 75 years (inclusive at both ends), only of Chinese ethnicity.
2. Patients with mature bones;
3. Patients with rotator cuff tear and/or shoulder joint instability requiring arthroscopic treatment;
4. Patients who are able to give voluntary and written informed consent to participate in the study and have signed EC-approved informed consent form.
5. Patients who are able to understand this clinical study, co-operates with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups for up to 12 months.

Exclusion Criteria:

1. Patients suffering from the rheumatic arthritis, tuberculosis of shoulder joint and infection around the shoulder joint;
2. Patients with massive rotator cuff tear that can't be repaired;
3. Patients who have received the rotator cuff surgery, arthroplasty of shoulder or surgical treatment of fracture for the shoulder joint at investigational side;
4. Patients with a bone defect existing in the glenoid cavity that need the reconstruction of bony defect in the glenoid cavity;
5. Patients that plan to receive the surgery for bilateral shoulder joint during the study;
6. Patients suffering from the bone diseases with pathological characteristics, such as cystic changes or severe osteoporosis, that may affect the safe fixation of anchor in the investigator's opinion;
7. Patients suffering from an active infection or sepsis (treated or untreated);
8. Patients suffering from other diseases (e.g. epilepsy) that may affect the results of shoulder joint function;
9. Patients that are known to be allergic to foreign body of materials of investigational product. If allergy to material is suspected, the corresponding test should be conducted and the possibility of allergy should be ruled out before implantation;
10. Patients suffering from serious cardiovascular disease, liver and kidney diseases;
11. Patients have an emotional or neurological condition that will affect their ability or willingness to participate in the study (e.g. cognitive disorder, mental illness, mental retardation).
12. Patients are immunosuppressed, have an autoimmune disorder, or an immune dysfunction. For examples, patients are on immunosuppressive therapy (cortisol at large dose, cytotoxic drugs, antilymphocytic serum or irradiation at large doses);
13. Patients are known to be at risk of being lost to follow-up, or failure to return to hospital for scheduled visits.
14. Patients participated in another clinical study of investigational drug, biologic, or device in the last 12 months.
15. Pregnant or lactating women, or those intend to become pregnant during the course of the study.
16. Known alcohol and/or drug abuse.
17. There are other serious or acute diseases, psychological conditions or social environment factors that may increase the risk of participating in the study or performing the surgery, or may reduce the reliability of participating in the study, or may increase the risk to the subjects themselves or others, in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female subjects
Enrollment: 128 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
The Constant-Murley score at 6 months after operation. | at 6 months after operation.
  Confirming Q-Fix is non-inferior to Twinfix, at 6 months after the repair of soft The Constant score is a 100 points scale consisting of four variables, which includes a patient reported part (pain 15 points and activity level 20 points), which results in a total of 35 points. Next to this there is a physician rated part (shoulder strength 25 points and range of motion 40 points) which totals 65 points.

CONTACTS AND LOCATIONS:
Overall Officials: Hui NA Yan, Doctor, Principal Investigator — Peking University Third Hospital
Locations (4):
- China (4):
  - Foshan Hospital of TCM, Foshan, Guangdong
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - 2nd Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Peking University Third Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No